CLINICAL TRIAL: NCT04760028
Title: Study on the Influencing Factors of Electroencephalogram Parameters Under Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EEG
Record Dates: First submitted 2021-02-05; First posted 2021-02-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: EEC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sevoflurane (Other): Adjust sevoflurane concentration as required
  Interventions: Procedure: Adjusting the depth of anesthesia

INTERVENTIONS:
Procedure: Adjusting the depth of anesthesia — After the main procedure, the depth of anesthesia can be adjusted as needed

SUMMARY:
The depth of anaesthesia is affected by the age factor in the interpretation of EEG information. Only by fully considering the influence of the age factor can we accurately grasp the depth of anaesthesia.

DETAILED DESCRIPTION:
In the process of general anesthesia, the reliable judgment of the depth of anesthesia has always been the focus of anesthesiologists.In recent decades, researchers have discovered that it is possible to monitor the effects of anesthesia using electroencephalography (EEG), so the information has come to be used to guide anesthesia management.The indicators derived from electroencephalogram (EEG) that can be used to judge the depth of anesthesia during general anesthesia, such as spectral edge frequency, burst inhibition rate, median power frequency, etc., were successively born. Thereafter, commercial instruments for monitoring the depth of anesthesia, such as EEG dual-frequency index, entropy module, Narcotrend index, etc., were also widely used in clinical practice.Although the anesthesia measurements or instrument has many advantages, but the use of these indicators are not considering the factors of age, and have been well documented for general anesthesia electroencephalography (eeg) of different ages is different, this means that in different age groups using the same monitoring indicators will lead to the judgment of anesthesia depth is larger error.Therefore, age should be considered in the process of monitoring the depth of clinical anesthesia, and appropriate indexes should be selected according to different ages to monitor the depth of anesthesia.However, it has not been thoroughly studied which indexes can be used to monitor the depth of anesthesia in each age group and how to conduct reasonable monitoring.Therefore, it is necessary to explore the monitoring indexes of depth of anesthesia in different age groups and the most appropriate monitoring program.

The purpose of this study was to validate EEG indicators that can monitor the depth of anesthesia at different ages, including basic EEG power spectrum parameters and processed parameters, and to explore whether there is an optimal protocol for monitoring the depth of anesthesia at different ages.In order to facilitate the clinical selection of patients of different age groups to monitor the depth of anesthesia, the factor of age is considered so as to take individual monitoring.Finally, it can accurately judge the depth of anesthesia and accurately use the anesthetic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅲ level
2. 18 to 100 years
3. BMI 19 ~ 30 kg/m squared
4. Patients without intracranial surgery

Exclusion Criteria:

1. nervous system diseases, abnormal EEG, old cerebral infarction, the use of drugs affecting the nervous system;
2. coronary heart disease, hypertension without regular treatment or poor control;
3. The oxygen partial pressure and calcium ion levels were abnormal before anesthesia induction;
4. History of alcohol abuse.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Indicators for monitoring the depth of anesthesia in different age groups | three months
  The absolute power of slow wave, δ wave, θ wave, α wave, β wave and γ wave in dB, the relative power of slow wave, δ wave, θ wave, α wave, β wave and γ wave in %, the approximate entropy, sequence entropy and sample entropy without unit, and the double coherence without unit in monitoring the depth of anesthesia in different ages
Relationship between EEG information index and age | three months
  The absolute power of slow wave, δ wave, θ wave, α wave, β wave and γ wave in dB, the relative power of slow wave, δ wave, θ wave, α wave, β wave and γ wave in %, there is no unit of approximate entropy, sequence entropy, sample entropy, double coherence and the relationship between age and depth of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Brown EN, Purdon PL. The aging brain and anesthesia. Curr Opin Anaesthesiol. 2013 Aug;26(4):414-9. doi: 10.1097/ACO.0b013e328362d183. PMID 23820102
- [Background] Bennett C, Voss LJ, Barnard JP, Sleigh JW. Practical use of the raw electroencephalogram waveform during general anesthesia: the art and science. Anesth Analg. 2009 Aug;109(2):539-50. doi: 10.1213/ane.0b013e3181a9fc38. PMID 19608830
- [Background] Otto KA, Cebotari S, Hoffler HK, Tudorache I. Electroencephalographic Narcotrend index, spectral edge frequency and median power frequency as guide to anaesthetic depth for cardiac surgery in laboratory sheep. Vet J. 2012 Mar;191(3):354-9. doi: 10.1016/j.tvjl.2011.02.023. Epub 2011 Mar 30. PMID 21454112
- [Background] Schultz A, Siedenberg M, Grouven U, Kneif T, Schultz B. Comparison of Narcotrend Index, Bispectral Index, spectral and entropy parameters during induction of propofol-remifentanil anaesthesia. J Clin Monit Comput. 2008 Apr;22(2):103-11. doi: 10.1007/s10877-008-9111-6. Epub 2008 Feb 21. PMID 18288579
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Hayashi K, Indo K, Sawa T. Anaesthesia-dependent oscillatory EEG features in the super-elderly. Clin Neurophysiol. 2020 Sep;131(9):2150-2157. doi: 10.1016/j.clinph.2020.05.027. Epub 2020 Jun 23. PMID 32682243
- [Background] Kreuzer M, Stern MA, Hight D, Berger S, Schneider G, Sleigh JW, Garcia PS. Spectral and Entropic Features Are Altered by Age in the Electroencephalogram in Patients under Sevoflurane Anesthesia. Anesthesiology. 2020 May;132(5):1003-1016. doi: 10.1097/ALN.0000000000003182. PMID 32108685
- [Background] Aranake A, Mashour GA, Avidan MS. Minimum alveolar concentration: ongoing relevance and clinical utility. Anaesthesia. 2013 May;68(5):512-22. doi: 10.1111/anae.12168. Epub 2013 Feb 16. PMID 23414556
- [Background] Blain-Moraes S, Tarnal V, Vanini G, Alexander A, Rosen D, Shortal B, Janke E, Mashour GA. Neurophysiological correlates of sevoflurane-induced unconsciousness. Anesthesiology. 2015 Feb;122(2):307-16. doi: 10.1097/ALN.0000000000000482. PMID 25296108
- [Background] Smith WD, Dutton RC, Smith NT. Measuring the performance of anesthetic depth indicators. Anesthesiology. 1996 Jan;84(1):38-51. doi: 10.1097/00000542-199601000-00005. PMID 8572353
- [Background] Li X, Li D, Liang Z, Voss LJ, Sleigh JW. Analysis of depth of anesthesia with Hilbert-Huang spectral entropy. Clin Neurophysiol. 2008 Nov;119(11):2465-75. doi: 10.1016/j.clinph.2008.08.006. Epub 2008 Sep 21. PMID 18812265